CLINICAL TRIAL: NCT04469153
Title: Interest of the Dosage of Ferritin / Glycosylated Ferritin in COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_FerriGly COVID
Record Dates: First submitted 2020-06-29; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: the Prognostic Value of Ferritin; Glycosylated Ferritin in SARS-CoV-2 Infection in Hospitalized COVID-19 Patients
Keywords: SARS-CoV-2; Ferritin; glycosylated ferritin; prognostic factor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-COV 2 positive patient: 57 SARS-COV-2 positive patients followed during the SARS-COV 2 epidemic in the internal medicine department of the Croix-Rousse hospital. For each patient ferritin and glycosylated ferritin was analysed one time (biological analysis) at the entry of the hospitalization.
  Interventions: Other: No intervention / Evaluation of the ferritin and glycosylated ferritin by standard approved serological tests

INTERVENTIONS:
Other: No intervention / Evaluation of the ferritin and glycosylated ferritin by standard approved serological tests — No intervention / Evaluation of the ferritin and glycosylated ferritin by standard approved serological tests

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a new coronavirus responsible for the pandemic called coronavirus disease 2019 (COVID-19), which appeared in China in December 2019 and which has spread rapidly around the world. Even if in the vast majority of viral infection results in a mild illness, it can also progress to a severe form with sometimes fatal consequences.

Indeed, clinical worsening, between the 7th and 10th days of the onset of symptoms, has been widely described since the start of the pandemic. This manifests itself at the biological level by hyperinflammation (VS, CRP, ferritin), coagulopathy (elevation of D-dimers, sometimes disseminated intravascular coagulation) and cell lysis (CPK, LDH).

At the same time, it was observed high levels of pro-inflammatory cytokines (IL-1β, IL-6, TNF-α, IL-18), suggestive of a cytokine storm, and the first studies on therapeutic management targeting these cytokines are currently underway in COVID-19.

Such a profile strongly recalls on the one hand the cytokine release syndrome (CRS, observed in CAR-T cell therapy in malignant hematology), and on the other hand the lymphohistiocytic activation syndrome (SALH). Systemic diseases, such as adult Still's disease and its pediatric side, can also be complicated by a cytokine storm, known as macrophagic activation syndrome (SAM, equivalent to secondary SALH). Under all these conditions, IL-1β, IL-18, IFN-γ and IL-6 seem to be key mediators of hyperinflammation.

Plasma ferritin is a biological marker of inflammation, long known, associated with various infectious, hematological and immunological conditions. An increase in ferritin levels has in particular been associated with an unfavorable development in certain infections such as influenza and certain authors have moreover shown an association between plasma ferritin and the evolution towards ARDS or death in patients. Its dosage is also used as a diagnostic tool for SAM, and could make it possible to differentiate the latter from severe sepsis in intensive care. Some authors have also noted it as a prognostic factor in Kawasaki disease or CRS.

The plasma dosage of ferritin, associated with that of its glycosylated fraction, could therefore be a diagnostic (difference between SAM and severe sepsis in intensive care), prognostic (evolution towards ARDS, mutation in intensive care, mortality) and therapeutic (indication of preemptive treatment with an inhibitor of IL-1 or IL6) in patients infected with SARS-CoV-2.

The objective of this study is to retrospectively assess the prognostic value of ferritin and glycosylated ferritin in SARS-CoV-2 infection in hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the internal medicine department of the Croix-Rousse hospital and positive for the SARS-COV 2 (nasopharyngeal sample, the test was appoved by the French national medical authorities).

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in the internal medicine department of the Croix-Rousse hospital and positive for the SARS-COV 2 (nasopharyngeal sample, the test was appoved by the French national medical authorities).
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
assessment of the prognostic value of ferritin in sars-cov2 positiv patients | the time point is measured one time (biological analysis) at the beginning of the hospitalization ie: day 0 (retrospective analysis).
  ferritin level will be assess by approved serological tests (French national medical authorities). Ferritin analysis is considered abnormal when the level is > at 388 µg/L;

CONTACTS AND LOCATIONS:
Locations (1):
- hopital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes, France